CLINICAL TRIAL: NCT04404712
Title: FAAH Availability in Psychiatric Disorders: A PET Study
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Ligand was not effective.
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Mohini Ranganathan, Associate Professor of Psychiatry, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2000027585
Record Dates: First submitted 2020-05-22; First posted 2020-05-27 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Post Traumatic Stress Disorder; Alcohol Use Disorder; Psychosis
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [11C]MK-3168 PET Scan (Experimental)
  Interventions: Drug: [11C]MK-3168

INTERVENTIONS:
Drug: [11C]MK-3168 — One PET scan involving administration of PET ligand [11C]MK-3168

SUMMARY:
The aim of the present study is to examine Fatty Acid Amide Hydrolase (FAAH) availability in humans, including healthy individuals and across a spectrum of psychiatric disorders in which alterations in the endocannabinoid system are observed.

DETAILED DESCRIPTION:
This study involves in vivo examination of FAAH availability, implicated both in the pathophysiology and therapeutics of disorders including PTSD, substance use disorders (e.g., alcohol use disorder, cannabis/cannabinoid use disorder, nicotine use disorder), psychotic disorders including schizophrenia, and mood disorders. The endocannabinoid system is a neuromodulatory system that has been implicated across a wide range of psychiatric disorders and may be implicated in the regulation of mood, appetitive behaviors, sleep, and cognition. Thus, alterations in the ECS have wide ranging implications. Finally, the ECS is being explored as a novel therapeutic target for several psychiatric disorders. Additionally, the test/retest reliability of the radiotracer, [11C]MK-3168, will be studied in up to 10 healthy control individuals.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65 years, inclusive
* Good physical health as determined by history, physical and laboratory examinations, ECG, and vital signs

PTSD Inclusion Criteria:

* Diagnosis of Post-Traumatic Stress Disorder

AUD Inclusion Criteria:

* Diagnosis of Alcohol Use Disorder

Psychosis Inclusion Criteria:

* Diagnosis of psychotic disorder such as Schizophrenia, Schizoaffective disorder

Exclusion Criteria:

* Presence of ferromagnetic metal in the body or heart pacemaker
* Women with a positive pregnancy test or women who are lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Total distribution of [11C]MK-3168 in the brain | PET scan day
  FAAH availability will be approximated using the FAAH positron emission tomography (PET) tracer [11C]MK-3168 total distribution

CONTACTS AND LOCATIONS:
Overall Officials: Mohini Ranganathan, MBBS, Principal Investigator — Neuroscience Research Training Program (NRTP); Office of Cooperative Research; Psychiatry; Schizophrenia Research Clinic; Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States